CLINICAL TRIAL: NCT03117660
Title: Effects of Retinoids on CYP2D6 Activity and Variability in Special Populations
Brief Title: Effects of Retinoids on CYP2D6 Activity During Pregnancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Mary Hebert, Professor of Pharmacy, Adjunct Professor of Obstetrics and Gynecology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001620; R01GM124264-01 (NIH)
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: CYP2D6 Polymorphism
MeSH Terms: interventions — Vitamin A

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, parallel group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin A (Experimental): Subjects will receive 3-4weeks of vitamin A
  Interventions: Drug: Vitamin A
- Control (No Intervention): Subjects will receive no treatment

INTERVENTIONS:
Drug: Vitamin A — vitamin A daily X3-4 weeks
  Arms: Vitamin A

SUMMARY:
Prospective drug interaction study during pregnancy.

DETAILED DESCRIPTION:
A randomized pharmacokinetic study to evaluate CYP2D6 activity with and without vitamin A administration during pregnancy and compared to postpartum control.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Extensive metabolizers

Exclusion Criteria:

* Chronic or persistent cough accompanying asthma, smoking or chronic obstructive pulmonary disease
* Productive cough
* Fever
* Known kidney disease
* Known liver disease
* Diabetes
* Obesity
* Bipolar disease
* Attention deficit disorder
* Social phobia
* Allergy or history of adverse event with dextromethorphan
* Drugs, foods, beverages or dietary supplements that interact with CYP2D6 or dextromethorphan
* dextromethorphan
* Unable to give written informed consent
* Inability to fast
* Concurrent use of vitamin A supplementation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy study
Enrollment: 82 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
CYP2D6 activity: dextromethorphan metabolic ratio | 4 weeks
  dextromethorphan metabolic ratio change from baseline during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Hebert, PharmD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will adhere to the NIH Grant Policy on Sharing Research Data. That is, after final data collection and analysis and after full peer review is performed on the data, the de-identified data generated by this project will be made available when requested by the academic community and researchers-at-large contingent upon Material Transfer Agreements with the University of Washington.

REFERENCES:
- [Background] Somani ST, Zeigler M, Fay EE, Leahy M, Bermudez B, Totah RA, Hebert MF. Changes in erythrocyte membrane epoxyeicosatrienoic, dihydroxyeicosatrienoic, and hydroxyeicosatetraenoic acids during pregnancy. Life Sci. 2021 Jan 1;264:118590. doi: 10.1016/j.lfs.2020.118590. Epub 2020 Oct 15. PMID 33069736
- [Background] Amaeze OU, Czuba LC, Yadav AS, Fay EE, LaFrance J, Shum S, Moreni SL, Mao J, Huang W, Isoherranen N, Hebert MF. Impact of Pregnancy and Vitamin A Supplementation on CYP2D6 Activity. J Clin Pharmacol. 2023 Mar;63(3):363-372. doi: 10.1002/jcph.2169. Epub 2022 Nov 15. PMID 36309846
- [Background] Czuba LC, Fay EE, LaFrance J, Smith CK, Shum S, Moreni SL, Mao J, Isoherranen N, Hebert MF. Plasma Retinoid Concentrations Are Altered in Pregnant Women. Nutrients. 2022 Mar 25;14(7):1365. doi: 10.3390/nu14071365. PMID 35405978